CLINICAL TRIAL: NCT07218068
Title: Intensive Preventative Dental Program Pilot Study
Acronym: IPDP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00082720; 03-21-01A (Other: Atrium Health)
Record Dates: First submitted 2025-10-15; First posted 2025-10-20 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-09

CONDITIONS: Dental Diseases
Keywords: Intensive Preventative Dental Program; dental caries; dental disease; prevention; head and neck cancer; Fluoride Varnishes; Osteoradionecrosis; dental infection
MeSH Terms: conditions — Stomatognathic Diseases; Dental Caries; Head and Neck Neoplasms; Osteoradionecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Intensive Preventative Dental Program (Experimental): head and neck cancer patients receive fluoride varnish applied to teeth and follow-up dental screening during regularly scheduled oncology appointments.
  Interventions: Drug: Fluoride varnish
- Regular Care (Active Comparator): control group consisting of head and neck cancer patients receiving regular care of no Intensive Preventative Dental Program.
  Interventions: Other: Regular Care
- Medical Oncology Team Providers (Experimental): Medical Oncology care team members (MD, DO, PA, NP, RN) who participate in Intensive Preventative Dental Program.
  Interventions: Other: Medical Oncology Care Team

INTERVENTIONS:
Drug: Fluoride varnish — fluoride varnish placed on teeth by a trained healthcare provider at four visits three months apart
  Arms: Intensive Preventative Dental Program
Other: Regular Care — standard oncology assessment visit without Intensive Preventative Dental Program services
  Arms: Regular Care
Other: Medical Oncology Care Team — Medical Oncology care team members participating in the Intensive Preventative Dental Program will be guided on recognizing dental disease and when it is appropriate to refer head and neck cancer patients for dental care.
  Arms: Medical Oncology Team Providers

SUMMARY:
Radiation therapy to treat cancer may cause a dry mouth from damage to salivary glands which may increase the risk of cavities on the teeth. The consistent use of prescription fluoride on teeth after radiation therapy for head and neck cancer may reduce the development of cavities and tooth loss. The purpose of this study is to find out if prescription fluoride varnish applied to the teeth every three months during the first year after radiation therapy changes the development of cavities or gum problems.

DETAILED DESCRIPTION:
The overall objective of this clinical trial is to determine if oncology practices can reduce dental disease in head and neck cancer patients post radiation therapy. Participants will have fluoride varnish applied at planned oncology follow-up visits and medical oncology providers will be instructed on recognizing dental disease and referring head and neck cancer patients for dental care when needed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* Willing and able to provide signed and dated consent form
* Presence of at least 4 natural erupted teeth remaining in the mouth after completion of pre-RT dental management
* Diagnosed with head and neck squamous cell carcinoma (SCC) or a salivary gland cancer (SGC), and intends to receive external beam radiation therapy (RT) with curative intent (tumor eradication), with or without concomitant chemotherapy;

OR

* Diagnosed with a non-SCC, non-SGC malignancy of the head and neck region, and intends to receive RT, with or without concomitant chemotherapy. The participant must be expected to receive at least 4500 cGy to one of the following sites:

  1. base of tongue
  2. buccal/labial mucosa
  3. epiglottis
  4. floor of mouth
  5. gingiva/alveolar ridge
  6. hard palate
  7. hypopharynx
  8. larynx
  9. lip
  10. mandible
  11. maxilla
  12. maxillary sinus
  13. nasal cavity
  14. nasopharynx
  15. neck
  16. oral cavity
  17. oral tongue
  18. oropharynx
  19. paranasal sinus/orbit
  20. parotid gland
  21. pharynx
  22. retromolar trigone
  23. soft palate
  24. sublingual gland
  25. submandibular gland
  26. tonsil;
* Willing to comply with all study procedures
* Willing to participate for the duration of the study
* RT follow-up planned for one of the selected AH Oncology Specialist Follow-up Sites.

Exclusion Criteria:

* Receiving palliative RT
* History of prior curative RT to the head and neck region to eradicate a malignancy.
* Incarcerated at the time of screening
* Anything that would place the participant at increased risk or preclude the participant's full compliance with or completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Change in Decayed, Missing and Filled Surfaces Score | from baseline to 12 months
  Decayed, Missing and Filled Surfaces Score (DMFS) is calculated by a calibrated oral examiner as the combined number of of decayed, missing, and/or filled tooth surfaces, from the baseline dental visit DMFS score before starting radiotherapy to the final dental visit DMFS score 12 months following completion of radiation therapy.

SECONDARY OUTCOMES:
Rate of Tooth Loss | from baseline to 12 months
  Number of teeth lost per participant as determined by a calculated oral examiner from the baseline dental visit before the start of radiotherapy to the dental visit 12 months after completing radiation therapy.
Rate of Oral Hygiene Compliance | from baseline to 12 months
  Number of participants who self-report daily toothbrushing and flossing from the baseline dental visit before the start of radiotherapy to the dental visit 12 months after completing radiation therapy.
Rate of Fluoride Compliance | from baseline to 12 months
  Number of participants who self-reported use of prescription fluoride daily from the baseline dental visit before the start of radiotherapy to the dental visit 12 months after completing radiation therapy.
Rate of Routine/Preventative Dental Care | from baseline to 12 months
  Number of participants who self-report visiting a dental office within the last six months from the baseline dental visit before the start of radiotherapy to the dental visit 12 months after completing radiation therapy.

OTHER OUTCOMES:
Medical Oncology Care Team Post-study Feasibility Survey | 12 months
  The feasibility survey evaluates the logistics and success in implementing the Intensive Preventative Dental Program for Medical Oncology Team Providers treating head and neck cancer patients by gathering feedback from the Medical Oncology Care Team. Items are scored with 1-5 point Likert scale with a lower scale indicating higher satisfaction with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Brennan, DDS, MHS, Principal Investigator — Atrium Health Wake Forest University Charlotte Medical Center; Matthew C. Ward, MD, Principal Investigator — Atrium Health Levine Cancer Center
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
As this is a pilot study which forms the basis of a larger clinical trial, individual deidentified participant data will be shared upon reasonable request to the primary investigators, along with a data dictionary outlining variables collected and data collection forms when appropriate.
Supporting Information: ICF
Time Frame: IPD will be available December 1, 2025 until at least December 1, 2030.
Access Criteria: Individual deidentified participant data as outlined above will be shared upon reasonable request to the primary investigators until the conclusion of the follow-up study (approximately December 2030)

DOCUMENTS (1):
  • Informed Consent Form (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/68/NCT07218068/ICF_000.pdf